CLINICAL TRIAL: NCT01786668
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study Of The Efficacy And Safety Of Tofacitinib In Subjects With Active Ankylosing Spondylitis (as)
Brief Title: Dose-Ranging Study Of Tofacitinib In Adults With Active Ankylosing Spondylitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921119; 2011-005689-39 (EudraCT Number)
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Results first posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-05

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; Spondylitis; Ankylosing; Spondyloarthritis; Spondyloarthropathy; Oral preparation
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylitis; Spondylarthritis; Spondylarthropathies | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Tofacitinib 2 mg (Experimental)
  Interventions: Drug: Tofacitinib 2 mg
- Tofacitinib 5 mg (Experimental)
  Interventions: Drug: Tofacitinib 5 mg
- Tofacitinib 10 mg (Experimental)
  Interventions: Drug: Tofacitinib 10 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tofacitinib 2 mg — 4 blinded tablets (two 1 mg tablets of tofacitinib along with two 5 mg matching placebo tablets) will be administered orally twice a day (in the AM and PM) for 12 weeks
  Arms: Tofacitinib 2 mg
Drug: Tofacitinib 5 mg — 4 blinded tablets (one 5 mg tablet of tofacitinib, one 5 mg and two 1 mg matching placebo tablets) will be administered orally twice a day (in the AM and PM) for 12 weeks
  Arms: Tofacitinib 5 mg
Drug: Tofacitinib 10 mg — 4 blinded tablets (two 5 mg tablets of tofacitinib and two 1 mg matching placebo tablets) will be administered orally twice a day (in the AM and PM) for 12 weeks
  Arms: Tofacitinib 10 mg
Drug: Placebo — 4 blinded tablets (two 1 mg and two 5 mg matching placebo tablets) will be administered orally twice a day (in the AM and PM) for 12 weeks
  Arms: Placebo

SUMMARY:
This is the first study of oral tofacitinib in adults with active ankylosing spondylitis. It is designed to obtain information on the efficacy and safety of 3 different doses of tofacitinib.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Ankylosing Spondylitis
* Has active disease despite concurrent nonsteroidal anti-inflammatory drugs (NSAIDs) treatment or is intolerant to NSAIDs

Exclusion Criteria:

* Pregnant or lactating females
* Currently receiving or previous use of a Tumor Necrosis Factor (TNF) inhibitor or any biological agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (67):
- United States (22):
  - Desert Medical Imaging, Indian Wells, California
  - Desert Medical Advances, Palm Desert, California
  - Arthritis & Rheumatology Associates, Clearwater, Florida
  - Millennium Research, Ormond Beach, Florida
  - Southwest Florida Clinical Research Center, Tampa, Florida
  - Covance Central Laboratory Services,Inc, Indianapolis, Indiana
  - Klein & Associates, M.D., P.A., Hagerstown, Maryland
  - Progressive Radiology, Hagerstown, Maryland
  - Advanced Medical Imaging (MRI center), Lincoln, Nebraska
  - Arthritis Center of Nebraska (X-ray center), Lincoln, Nebraska
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Charlotte Radiology/ Carolina Imaging Services, Ballantyne, North Carolina
  - Joint and Muscle Research Institute, Charlotte, North Carolina
  - Presbyterian Imaging, Charlotte, North Carolina
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - Premier Physicians Centers, Westlake, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, LLC, Wyomissing, Pennsylvania
  - Investigational Drug Service, Seatle, Washington
  - Seattle Rheumatology Associates, Seattle, Washington
  - Arthritis Northwest, PLLC, Spokane, Washington
- Canada (2):
  - Institut de Rhumatologie de Montreal, Montreal, Quebec
  - G.R.M.O. Inc, Québec, Quebec
- Czechia (5):
  - Artroscan s.r.o., Ostrava, Czech Republic
  - Revmatologicky ustav, Prague
  - Revmatologicka ambulance, Prague
  - Mediscan Group s.r.o., Praha 11- Chodov
  - Medical Plus, Uherské Hradiště
- Germany (4):
  - Charité Universitaetsmedizin Berlin, Berlin
  - Praxis fuer klinische Studien, Hamburg
  - Gemeinschaftspraxis Dres. von Hinueber / Demary, Hildesheim
  - Immunologisches Zentrum Vogelsang-Gommern GmbH, Vogelsang-Gommern
- Hungary (7):
  - Dr. Rethy Pál Korhaz es Rendelointezet, Reumatologia, Békéscsaba
  - Orszagos Reumatologiai es Fiziotherapias Intezet II. Reumatologiai Osztaly, Budapest
  - Qualiclinic Kft, Budapest
  - Synexus Magyarorszag Kft. - Synexus Hungary Clinical Research Centre, Budapest
  - Debreceni Egyetem Orvos- és Egészségtudományi Centrum, Debrecen
  - CRU Hungary Kft., Szikszó
  - Csolnoky Ferenc Korhaz Reumatologiai Osztaly, Veszprém
- Poland (9):
  - NZOZ Lecznica MAK-MED s.c., Nadarzyn, Masovian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej Centrum Osteoporozy i Chorob Kostno-Stawowych, Bialystok
  - Szpital Uniwersytecki nr 2 im. dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Kliniczno-Badawcze J. Brzezicki, B. Gornikiewicz-Brzezicka Lekarze Spolka Partnerska, Elblag
  - Medica Pro Familia Sp. z o.o. S.K.A. Oddzial Katowice, Katowice
  - Malopolskie Centrum Medyczne S.C., Krakow
  - Zespol Poradni Specjalistycznych Reumed Filia Onyksowa, Lublin
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól
  - NZOZ Nasz Lekarz Praktyka Grupowa Lekarzy Rodzinnych z Przychodnia Specjalistyczna w Toruniu, Torun
- Russia (4):
  - Federal State Budgetary Institution, Moscow
  - OOO AVA-PETER "Scandinavia clinic", Saint Petersburg
  - Saint-Petersburg State Budgetary Healthcare Institution, Sestroretsk
  - SBEI HPE Ural State Medical University of MoH of RF based on Municipal Budgetary Institution, Yekaterinburg
- South Korea (4):
  - Chonnam National University Hospital, Gwangju
  - INHA University Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (7):
  - Complexo Hospitalario Universitario A Coruna, A Coruña, A Coruna
  - Hospital Clinico Universitario Santiago de Compostela, Santiago de Compostela, A Coruna
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - Hospital Universitario De La Paz, Madrid
  - Corporacio Sanitaria Parc Tauli, Sabadell
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - China medical university hospital, Taichung

REFERENCES:
- [Derived] Deodhar A, Akar S, Curtis JR, El-Zorkany B, Magrey M, Wang C, Wu J, Makgoeng SB, Vranic I, Menon S, Fleishaker DL, Diehl AM, Fallon L, Yndestad A, Landewe RBM. Integrated safety analysis of tofacitinib from Phase 2 and 3 trials of patients with ankylosing spondylitis. Adv Rheumatol. 2024 Dec 18;64(1):87. doi: 10.1186/s42358-024-00402-x. PMID 39695887
- [Derived] Norton H, Sliwinska-Stanczyk P, Hala T, El-Zorkany B, Stockert L, Mundayat R, Wang L, Ritchlin CT. Tofacitinib Efficacy/Safety in Patients with Ankylosing Spondylitis by Baseline Body Mass Index: A Post Hoc Analysis of Phase 2/3 Trials. Rheumatol Ther. 2025 Feb;12(1):67-84. doi: 10.1007/s40744-024-00726-6. Epub 2024 Dec 5. PMID 39636343
- [Derived] Deodhar A, Baraliakos X, Magrey M, Gensler LS, Thorat AV, Pemmaraju SK, Cadatal MJ, Nash P. Efficacy and Safety of Tofacitinib in Ankylosing Spondylitis by Baseline C-Reactive Protein Level: Post Hoc Analysis of Phase II and Phase III Clinical Trials. J Rheumatol. 2024 Aug 1;51(8):772-780. doi: 10.3899/jrheum.2023-1198. PMID 38825359
- [Derived] Kristensen LE, Deodhar A, Leung YY, Vranic I, Mortezavi M, Fallon L, Yndestad A, Kinch CD, Gladman DD. Risk Stratification of Patients with Psoriatic Arthritis and Ankylosing Spondylitis for Treatment with Tofacitinib: A Review of Current Clinical Data. Rheumatol Ther. 2024 Jun;11(3):487-499. doi: 10.1007/s40744-024-00662-5. Epub 2024 May 2. PMID 38696034
- [Derived] Magrey M, Wei JC, Yndestad A, Bushmakin AG, Cappelleri JC, Dina O, Deodhar A. Relationships of Work Productivity and Activity Impairment With Patient-Reported Outcomes in Ankylosing Spondylitis: Results From Two Trials. Arthritis Care Res (Hoboken). 2024 Mar;76(3):359-365. doi: 10.1002/acr.25267. Epub 2024 Jan 5. PMID 37909386
- [Derived] Ostergaard M, Wu J, Fallon L, Sherlock SP, Wang C, Fleishaker D, Kanik KS, Maksymowych WP. Tofacitinib Reduces Spinal Inflammation in Vertebral Bodies and Posterolateral Elements in Ankylosing Spondylitis: Results from a Phase 2 Trial. Rheumatol Ther. 2023 Aug;10(4):1001-1020. doi: 10.1007/s40744-023-00564-y. Epub 2023 Jun 18. PMID 37331992
- [Derived] Cella D, Lenderking WR, Chongpinitchai P, Bushmakin AG, Dina O, Wang L, Cappelleri JC, Navarro-Compan V. Functional Assessment of Chronic Illness Therapy-Fatigue is a reliable and valid measure in patients with active ankylosing spondylitis. J Patient Rep Outcomes. 2022 Sep 23;6(1):100. doi: 10.1186/s41687-022-00508-0. PMID 36138330
- [Derived] van der Heijde D, Deodhar A, Wei JC, Drescher E, Fleishaker D, Hendrikx T, Li D, Menon S, Kanik KS. Tofacitinib in patients with ankylosing spondylitis: a phase II, 16-week, randomised, placebo-controlled, dose-ranging study. Ann Rheum Dis. 2017 Aug;76(8):1340-1347. doi: 10.1136/annrheumdis-2016-210322. Epub 2017 Jan 27. PMID 28130206
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921119&StudyName=Dose-Ranging%20Study%20Of%20Tofacitinib%20In%20Adults%20With%20Active%20Ankylosing%20Spondylitis

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total 208 participants were randomized to double-blind treatment; 52 to each treatment group (tofacitinib 2 milligrams [mg] twice daily [BID], tofacitinib 5 mg BID, tofacitinib 10 mg BID, and placebo BID). One participant was randomized to the placebo group but did not receive study drug, as such only 207 participants received study treatment.
Groups:
- Tofacitinib 2 mg BID: Participants were administered 4 tablets (two 1 mg tablets of tofacitinib along with two 5 mg matching placebo tablets) orally BID (in the morning [AM] and afternoon [PM]) for a total of 12 weeks.
- Tofacitinib 5 mg BID: Participants were administered 4 tablets (one 5 mg tablet of tofacitinib, one 5 mg and two 1 mg matching placebo tablets) orally BID (in the AM and PM) for a total of 12 weeks.
- Tofacitinib 10 mg BID: Participants were administered 4 tablets (two 5 mg tablets of tofacitinib and two 1 mg matching placebo tablets) orally twice a day (in the AM and PM) for a total of 12 weeks.
- Placebo BID: Participants were administered 4 tablets (two 1 mg placebo tablets and two 5 mg matching placebo tablets) orally twice a day (in the AM and PM) for a total of 12 weeks.
Period: Overall Study
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Started | 52 | 52 | 52 | 51
Completed | 51 | 51 | 47 | 47
Not Completed | 1 | 1 | 5 | 4
Not completed — Adverse Event | 0 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population - included participants who received at least 1 dose of study medication
Groups:
- Tofacitinib 2 mg BID: Participants were administered 4 tablets (two 1 mg tablets of tofacitinib along with two 5 mg matching placebo tablets) orally BID (in the AM and PM) for a total of 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID | Total
Number analyzed (Participants) | 52 | 52 | 52 | 51 | 207
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age | 41.8 (12.3) | 41.2 (10.3) | 41.6 (12.2) | 41.9 (12.9) | 41.6 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 14 | 19 | 64
  Male | 34 | 39 | 38 | 32 | 143

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving 20 Percent (%) Improvement in Assessment of SpondyloArthritis International Society (ASAS) Score (ASAS 20) at Week 12
Description: The primary analysis of this outcome measure was performed using the Emax model. Clinical response to treatment was assessed according to ASAS20 criteria. ASAS20 responder had improvement of greater than or equal to (≥) 20% and ≥1 unit in at least 3 domains (on a scale of 0 [least] to 10 [worst]) and no worsening of ≥20% and less than or equal to (≤)1 unit in the remaining domain. The domains are: Patient's Global Assessment of Disease Activity, spinal pain, function and inflammation (from Bath Ankylosing Spondylitis Disease Activity Index [BASDAI]). Missing data were handled by nonresponsive (NRI)/ last observation carried forward (LOCF). Missing values due to a subject dropping out from the study were handled by setting the ASAS20 value to NRI. The LOCF approach was applied to missing components, if just some of the components of the ASAS20 were missing.
Time Frame: Week 12
Population: Full Analysis Set (FAS): included all participants who were randomized to the study and received at least one dose of the randomized study drug (Tofacitinib or placebo).
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 52 | 52 | 52 | 51
Percentage of participants | 56.0 | 63.0 | 67.4 | 40.1
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Emax model - 95% Confidence Interval represents 95% Credible Interval; Test type: Superiority or Other; Emax Model; Risk Difference (RD) = 15.8, 95% CI 2-sided [5.0 to 30.3]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Emax model - 95% Confidence Interval represents 95% Credible Interval; Test type: Superiority or Other; Emax Model; Risk Difference (RD) = 22.9, 95% CI 2-sided [8.4 to 37.7]
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Emax model - 95% Confidence Interval represents 95% Credible Interval; Test type: Superiority or Other; Emax Model; Risk Difference (RD) = 27.3, 95% CI 2-sided [10.7 to 43.4]

2. Primary Outcome: Percentage of Participants Achieving ASAS20 at Week 12
Description: The supportive analysis of this outcome measure was performed using the normal approximation for two proportions. Clinical response to treatment was assessed according to ASAS20 criteria. ASAS20 responder had improvement of ≥ 20% and ≥1 unit in at least 3 domains (on a scale of 0 [least] to 10 [worst]) and no worsening of ≥20% and ≤1 unit in the remaining domain. The domains are: Patient's Global Assessment of Disease Activity, spinal pain, function and inflammation (from Bath Ankylosing Spondylitis Disease Activity Index [BASDAI]). Missing data were handled by NRI/LOCF. Missing values due to a subject dropping out from the study were handled by setting the ASAS20 value to NRI. The LOCF approach was applied to missing components, if just some of the components of the ASAS20 were missing.
Time Frame: Baseline, Week 12
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 52 | 52 | 52 | 51
Percentage of participants | 51.92 | 80.77 | 55.77 | 41.18
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.271, Normal approximation for two proportions; Risk Difference (RD) = 10.75, 95% CI 2-sided [-8.41 to 29.90], Standard Error of Mean 9.77
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.001, Normal approximation for two proportions; Risk Difference (RD) = 39.59, 95% CI 2-sided [22.35 to 56.83], Standard Error of Mean 8.80
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.134, Normal approximation for two proportions; Risk Difference (RD) = 14.59, 95% CI 2-sided [-4.50 to 33.69], Standard Error of Mean 9.74

3. Secondary Outcome: Percentage of Participants Achieving 20% Improvement in ASAS Score at Weeks 2, 4 and 8
Description: Clinical response to treatment was assessed according to ASAS20 criteria. ASAS20 responder had improvement of ≥ 20% and ≥1 unit in at least 3 domains (on a scale of 0 [least] to 10 [worst]) and no worsening of ≥20% and ≤1 unit in the remaining domain. The domains are: Patient's Global Assessment of Disease Activity, spinal pain, function and inflammation (from Bath Ankylosing Spondylitis Disease Activity Index [BASDAI]). Missing data were handled by NRI/LOCF. Missing values due to a subject dropping out from the study were handled by setting the ASAS20 value to NRI. The LOCF approach was applied to missing components, if just some of the components of the ASAS20 were missing.
Time Frame: Baseline, Week 2, Week 4, Week 8
Population: FAS - n=number of responders at each visit.
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 52 | 52 | 52 | 51
Percentage of participants
  Week 2 (n=21,17,18,14) | 40.38 | 32.69 | 34.62 | 27.45
  Week 4 (n=25,29,25,17) | 48.08 | 55.77 | 48.08 | 33.33
  Week 8 (n=30, 37, 28, 22) | 57.69 | 71.15 | 53.85 | 43.14
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.162, Normal approximation for two proportions; Risk Difference (RD) = 12.93, 95% CI 2-sided [-5.17 to 31.04], Standard Error of Mean 9.24
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.561, Normal approximation for two proportions; Risk Difference (RD) = 5.24, 95% CI 2-sided [-12.44 to 22.92], Standard Error of Mean 9.02
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.430, Normal approximation for two proportions; Risk Difference (RD) = 7.16, 95% CI 2-sided [-10.65 to 24.97], Standard Error of Mean 9.09
Statistical Analysis 4: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.123, Normal approximation for two proportions; Risk Difference (RD) = 14.74, 95% CI 2-sided [-4.01 to 33.50], Standard Error of Mean 9.57
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.019, Normal approximation for two proportions; Risk Difference (RD) = 22.44, 95% CI 2-sided [3.74 to 41.13], Standard Error of Mean 9.54
Statistical Analysis 6: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.123, Normal approximation for two proportions; Risk Difference (RD) = 14.74, 95% CI 2-sided [-4.01 to 33.50], Standard Error of Mean 9.57
Statistical Analysis 7: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.135, Normal approximation for two proportions; Risk Difference (RD) = 14.56, 95% CI 2-sided [-4.55 to 33.66], Standard Error of Mean 9.75
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.003, Normal approximation for two proportions; Risk Difference (RD) = 28.02, 95% CI 2-sided [9.68 to 46.36], Standard Error of Mean 9.36
Statistical Analysis 9: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.274, Normal approximation for two proportions; Risk Difference (RD) = 10.71, 95% CI 2-sided [-8.48 to 29.90], Standard Error of Mean 9.79

4. Secondary Outcome: Change From Baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) Magnetic Resonance Imaging (MRI) Index of Disease Activity Score of the Sacroiliac (SI) Joints at Week 12
Description: SPARCC scoring consists of assessing six SI joint MRI image coronal slices representing the largest proportion of the synovial compartment of the SI joints for edema. The maximum score per slice was 2 and 12 for all 6 slices. The total minimum and maximum score for all SI joints across 6 slices is 0 to 72 and higher scores indicate more inflammation. A negative change from baseline indicates improvement. Missing data at Week 12 were imputed by LOCF if data at an early visit (discontinuation visit) were available.
Time Frame: Baseline, Week 12
Population: FAS - when change from baseline is analyzed, FAS requires that participants have a baseline and at least one post-baseline measurement
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 42 | 44 | 44 | 34
Units on a scale | -1.70 (0.779) | -3.15 (0.788) | -3.55 (0.795) | -0.81 (0.806)
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.427, ANCOVA; Mean Difference (Final Values) = -0.89, 95% CI 2-sided [-3.11 to 1.32], Standard Error of Mean 1.123
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.039, ANCOVA; Mean Difference (Final Values) = -2.35, 95% CI 2-sided [-4.58 to -0.12], Standard Error of Mean 1.130
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.016, ANCOVA; Mean Difference (Final Values) = -2.74, 95% CI 2-sided [-4.97 to -0.51], Standard Error of Mean 1.131

5. Secondary Outcome: Change From Baseline in SPARCC MRI Index of Disease Activity Score of the Spine at Week 12
Description: SPARCC scoring of the magnetic resonance imaging (MRI) of the spine consists of assessing six disco-vertebral units (DVU) with 3 consecutive sagittal slices at each DVU. The minimum and maximum SPARCC score for all 6 DVUs is 0 to 108, with higher scores indicating more damage. A negative change from baseline indicates improvement. Missing data at Week 12 were imputed by LOCF if data at an early visit (discontinuation visit) were available.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 41 | 44 | 44 | 34
Units on a scale | -3.09 (1.061) | -5.51 (1.063) | -6.57 (1.073) | -0.09 (1.085)
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.050, ANCOVA; Mean Difference (Final Values) = -3.00, 95% CI 2-sided [-5.99 to -0.00], Standard Error of Mean 1.517
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -5.42, 95% CI 2-sided [-8.42 to -2.42], Standard Error of Mean 1.520
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -6.47, 95% CI 2-sided [-9.48 to -3.46], Standard Error of Mean 1.525

6. Secondary Outcome: Change From Baseline in Modified Berlin Ankylosing Spondylitis Spine Magnetic Resonance Imaging Activity Score (ASspiMRI) of the Spine at Week 12
Description: Berlin modification of the ASspiMRI is a measure of acute lesion as determined by short-tau inversion recovery (STIR) sequences. All 23 disco-vertebral units (DVU) of the spine (from C2 to S1), defined as the region between 2 virtual lines through the middle of each vertebra, were scored in a single dimension, which is represented the highest level of inflammation in that particular DVU. Total spine ASspiMRI scores can range from 0-69 with higher scores indicating more disease activity. A negative change from baseline indicates improvement. Missing data at Week 12 were imputed by LOCF if data at an early visit (discontinuation visit) were available.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 41 | 44 | 44 | 34
Units on a scale | -1.05 (0.364) | -2.22 (0.364) | -2.13 (0.368) | -0.41 (0.372)
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.221, ANCOVA; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-1.66 to 0.39], Standard Error of Mean 0.520
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.80, 95% CI 2-sided [-2.83 to -0.78], Standard Error of Mean 0.520
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = -1.71, 95% CI 2-sided [-2.75 to -0.68], Standard Error of Mean 0.523

7. Secondary Outcome: Percentage of Participants Achieving 40% Improvement in ASAS Score at Weeks 2, 4, 8 and 12
Description: ASAS 40 is defined as ≥40% and absolute change of ≥2 units in at least 3 domains on a 0-10 scale (0=no disease activity, 10=high disease activity), and no worsening in the remaining domain. Missing data were handled by NRI/LOCF.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: FAS - n=number of responders at each visit.
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 52 | 52 | 52 | 51
Percentage of participants
  Week 2 (n=7, 7, 9, 8) | 13.46 | 13.46 | 17.31 | 15.69
  Week 4 (n=15, 17, 11, 8) | 28.85 | 32.69 | 21.15 | 15.69
  Week 8 (n=15, 18, 19, 14) | 28.85 | 34.62 | 36.54 | 27.45
  Week 12 (n=22, 24, 20, 10) | 42.31 | 46.15 | 38.46 | 19.61
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.749, Normal approximation for two proportions; Risk Difference (RD) = -2.22, 95% CI 2-sided [-15.85 to 11.40], Standard Error of Mean 6.95
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.749, Normal approximation for two proportions; Risk Difference (RD) = -2.22, 95% CI 2-sided [-15.85 to 11.40], Standard Error of Mean 6.95
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.824, Normal approximation for two proportions; Risk Difference (RD) = 1.62, 95% CI 2-sided [-12.71 to 15.95], Standard Error of Mean 7.31
Statistical Analysis 4: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.104, Normal approximation for two proportions; Risk Difference (RD) = 13.16, 95% CI 2-sided [-2.69 to 29.01], Standard Error of Mean 8.09
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.040, Normal approximation for two proportions; Risk Difference (RD) = 17.01, 95% CI 2-sided [0.81 to 33.20], Standard Error of Mean 8.26
Statistical Analysis 6: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.473, Normal approximation for two proportions; Risk Difference (RD) = 5.47, 95% CI 2-sided [-9.46 to 20.40], Standard Error of Mean 7.62
Statistical Analysis 7: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.875, Normal approximation for two proportions; Risk Difference (RD) = 1.40, 95% CI 2-sided [-15.97 to 18.76], Standard Error of Mean 8.86
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.430, Normal approximation for two proportions; Risk Difference (RD) = 7.16, 95% CI 2-sided [-10.65 to 24.97], Standard Error of Mean 9.09
Statistical Analysis 9: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.320, Normal approximation for two proportions; Risk Difference (RD) = 9.09, 95% CI 2-sided [-8.84 to 27.01], Standard Error of Mean 9.15
Statistical Analysis 10: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.010, Normal approximation for two proportions; Risk Difference (RD) = 22.70, 95% CI 2-sided [5.41 to 39.99], Standard Error of Mean 8.82
Statistical Analysis 11: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.003, Normal approximation for two proportions; Risk Difference (RD) = 26.55, 95% CI 2-sided [9.16 to 43.93], Standard Error of Mean 8.87
Statistical Analysis 12: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.031, Normal approximation for two proportions; Risk Difference (RD) = 18.85, 95% CI 2-sided [1.72 to 35.99], Standard Error of Mean 8.74

8. Secondary Outcome: Percentage of Participants Achieving ASAS5/6 Response at Weeks 2, 4, 8 and 12
Description: ASAS5/6 consists of 6 domains: the 4 used in ASAS20 (Patient's Global Assessment of Disease Activity, spinal pain, function, inflammation plus spinal mobility and an acute phase reactant, C Reactive Protein (CRP). ASAS 5/6 is defined as ≥20% improvement in at least 5 domains and no worsening in the remaining domain. Missing data were handled by NRI/LOCF.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: FAS - n=number of responders at each visit
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 52 | 52 | 52 | 51
Percentage of participants
  Week 2 (n=12, 7, 11, 4) | 23.08 | 13.46 | 21.15 | 7.84
  Week 4 (n=10, 16, 15, 4) | 19.23 | 30.77 | 28.85 | 7.84
  Week 8 (n=11, 22, 15, 5) | 21.15 | 42.31 | 28.85 | 9.80
  Week 12 (n=10, 26, 20, 8) | 19.23 | 50.00 | 38.46 | 15.69
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.028, Normal approximation for two proportions; Risk Difference (RD) = 15.23, 95% CI 2-sided [1.61 to 28.86], Standard Error of Mean 6.95
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.353, Normal approximation for two proportions; Risk Difference (RD) = 5.62, 95% CI 2-sided [-6.23 to 17.47], Standard Error of Mean 6.05
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.050, Normal approximation for two proportions; Risk Difference (RD) = 13.31, 95% CI 2-sided [-0.02 to 26.64], Standard Error of Mean 6.80
Statistical Analysis 4: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.086, Normal approximation for two proportions; Risk Difference (RD) = 11.39, 95% CI 2-sided [-1.62 to 24.39], Standard Error of Mean 6.64
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.002, Normal approximation for two proportions; Risk Difference (RD) = 22.93, 95% CI 2-sided [8.37 to 37.48], Standard Error of Mean 7.43
Statistical Analysis 6: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.004, Normal approximation for two proportions; Risk Difference (RD) = 21.00, 95% CI 2-sided [6.65 to 35.36], Standard Error of Mean 7.32
Statistical Analysis 7: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.106, Normal approximation for two proportions; Risk Difference (RD) = 11.35, 95% CI 2-sided [-2.43 to 25.13], Standard Error of Mean 7.03
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p < 0.001, Normal approximation for two proportions; Risk Difference (RD) = 32.50, 95% CI 2-sided [16.79 to 48.22], Standard Error of Mean 8.02
Statistical Analysis 9: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.012, Normal approximation for two proportions; Risk Difference (RD) = 19.04, 95% CI 2-sided [4.27 to 33.81], Standard Error of Mean 7.54
Statistical Analysis 10: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.635, Normal approximation for two proportions; Risk Difference (RD) = 3.54, 95% CI 2-sided [-11.10 to 18.19], Standard Error of Mean 7.47
Statistical Analysis 11: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p < 0.001, Normal approximation for two proportions; Risk Difference (RD) = 34.31, 95% CI 2-sided [17.45 to 51.18], Standard Error of Mean 8.60
Statistical Analysis 12: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.007, Normal approximation for two proportions; Risk Difference (RD) = 22.78, 95% CI 2-sided [6.21 to 39.34], Standard Error of Mean 8.45

9. Secondary Outcome: Change From Baseline of Ankylosing Spondylitis Disease Activity Score Using C-Reactive Protein ASDAS(CRP) at Weeks 2, 4, 8 and 12
Description: The ASDAS(CRP) is a derived score that uses back pain, duration of morning stiffness, Patient's Global Assessment of their disease and peripheral pain/swelling. The formula used for calculating the ASDAS (CRP)is: 0.12 x Back Pain + 0.06 x Duration of Morning Stiffness + 0.11 x Patient Global + 0.07 x Peripheral Pain/Swelling + 0.58 x Ln(CRP+1). The calculated score can be from 0 to no defined upper limit. A negative number indicates a reduction in the score which indicates decrease in disease activity.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 51 | 51 | 51 | 50
Units on a scale
  Week 2 | -0.68 (0.096) [15.20 to 39.70] | -1.00 (0.096) | -0.97 (0.096) | -0.50 (0.097)
  Week 4 | -1.01 (0.099) | -1.20 (0.099) | -1.17 (0.099) | -0.58 (0.100)
  Week 8 | -1.08 (0.111) | -1.36 (0.111) | -1.32 (0.112) | -0.73 (0.112)
  Week 12 | -1.23 (0.119) | -1.41 (0.119) | -1.37 (0.121) | -0.68 (0.123)
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.175, Mixed Models Analysis; Includes fixed effects of treatment group, visit, and treatment-group by-visit interaction and baseline value, using an unstructured covariance matrix; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.46 to 0.08], Standard Error of Mean 0.136
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-0.77 to -0.24], Standard Error of Mean 0.136
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.74 to -0.20], Standard Error of Mean 0.136
Statistical Analysis 4: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-0.70 to -0.15], Standard Error of Mean 0.141
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-0.90 to -0.34], Standard Error of Mean 0.141
Statistical Analysis 6: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-0.86 to -0.31], Standard Error of Mean 0.141
Statistical Analysis 7: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.026, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.66 to -0.04], Standard Error of Mean 0.158
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-0.94 to -0.32], Standard Error of Mean 0.157
Statistical Analysis 9: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-0.90 to -0.27], Standard Error of Mean 0.159
Statistical Analysis 10: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.89 to -0.21], Standard Error of Mean 0.171
Statistical Analysis 11: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.73, 95% CI 2-sided [-1.07 to -0.39], Standard Error of Mean 0.171
Statistical Analysis 12: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-1.03 to -0.35], Standard Error of Mean 0.172

10. Secondary Outcome: Percentage of Participants With ASDAS Clinically Important Improvement at Weeks 2, 4, 8 and 12
Description: The ASDAS clinically important improvement was calculated from the ASDAS data. The ASDAS clinically important improvement is defined as change (decrease) from baseline of ≥1.1 units. Missing data were handled by NRI/LOCF.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: FAS - n=number of responders at each visit
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 52 | 52 | 52 | 51
Percentage of participants
  Week 2 (n=14, 25, 21, 8) | 26.92 | 48.08 | 40.38 | 15.69
  Week4 (n=22, 30, 27, 10) | 42.31 | 57.69 | 51.92 | 19.61
  Week 8 (n=23, 31, 31, 15) | 44.23 | 59.62 | 59.62 | 29.41
  Week 12 (n=27, 33, 29, 14) | 51.92 | 63.46 | 55.77 | 27.45
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.159, Normal approximation for two proportions; Risk Difference (RD) = 11.24, 95% CI 2-sided [-4.41 to 26.89], Standard Error of Mean 7.99
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p < 0.001, Normal approximation for two proportions; Risk Difference (RD) = 32.39, 95% CI 2-sided [15.54 to 49.24], Standard Error of Mean 8.60
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.004, Normal approximation for two proportions; Risk Difference (RD) = 24.70, 95% CI 2-sided [8.04 to 41.36], Standard Error of Mean 8.50
Statistical Analysis 4: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.010, Normal approximation for two proportions; Risk Difference (RD) = 22.70, 95% CI 2-sided [5.41 to 39.99], Standard Error of Mean 8.82
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p < 0.001, Normal approximation for two proportions; Risk Difference (RD) = 38.08, 95% CI 2-sided [20.79 to 55.38], Standard Error of Mean 8.82
Statistical Analysis 6: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p < 0.001, Normal approximation for two proportions; Risk Difference (RD) = 32.32, 95% CI 2-sided [14.90 to 49.73], Standard Error of Mean 8.88
Statistical Analysis 7: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.114, Normal approximation for two proportions; Risk Difference (RD) = 14.82, 95% CI 2-sided [-3.58 to 33.22], Standard Error of Mean 9.39
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.001, Normal approximation for two proportions; Risk Difference (RD) = 30.20, 95% CI 2-sided [11.92 to 48.49], Standard Error of Mean 9.33
Statistical Analysis 9: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.001, Normal approximation for two proportions; Risk Difference (RD) = 30.20, 95% CI 2-sided [11.92 to 48.49], Standard Error of Mean 9.33
Statistical Analysis 10: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.009, Normal approximation for two proportions; Risk Difference (RD) = 24.47, 95% CI 2-sided [6.18 to 42.76], Standard Error of Mean 9.33
Statistical Analysis 11: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p < 0.001, Normal approximation for two proportions; Risk Difference (RD) = 36.01, 95% CI 2-sided [18.09 to 53.94], Standard Error of Mean 9.15
Statistical Analysis 12: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.002, Normal approximation for two proportions; Risk Difference (RD) = 28.32, 95% CI 2-sided [10.09 to 46.55], Standard Error of Mean 9.30

11. Secondary Outcome: Percentage of Participants With ASDAS Major Improvement at Weeks 2, 4, 8 and 12
Description: The ASDAS major improvement was calculated from the ASDAS data. The ASDAS major improvement was defined as change (decrease) from baseline of ≥2.0 units. Missing data were handled by NRI/LOCF.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: FAS - n=number of responders at each visit
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 52 | 52 | 52 | 51
Percentage of participants
  Week 2 (n=4, 4, 4, 1) | 7.69 | 7.69 | 7.69 | 1.96
  Week 4 (n=6, 6, 8, 3) | 11.54 | 11.54 | 15.38 | 5.88
  Week 8 (n=6, 14, 12, 5) | 11.54 | 26.92 | 23.08 | 9.80
  Week 12 (n=10, 12, 13, 6) | 19.23 | 23.08 | 25.00 | 11.76
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.170, Normal approximation for two proportions; Risk Difference (RD) = 5.73, 95% CI 2-sided [-2.45 to 13.91], Standard Error of Mean 4.17
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.170, Normal approximation for two proportions; Risk Difference (RD) = 5.73, 95% CI 2-sided [-2.45 to 13.91], Standard Error of Mean 4.17
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.170, Normal approximation for two proportions; Risk Difference (RD) = 5.73, 95% CI 2-sided [-2.45 to 13.91], Standard Error of Mean 4.17
Statistical Analysis 4: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.306, Normal approximation for two proportions; Risk Difference (RD) = 5.66, 95% CI 2-sided [-5.17 to 16.48], Standard Error of Mean 5.52
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.306, Normal approximation for two proportions; Risk Difference (RD) = 5.66, 95% CI 2-sided [-5.17 to 16.48], Standard Error of Mean 5.52
Statistical Analysis 6: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.113, Normal approximation for two proportions; Risk Difference (RD) = 9.50, 95% CI 2-sided [-2.24 to 21.24], Standard Error of Mean 5.99
Statistical Analysis 7: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.775, Normal approximation for two proportions; Risk Difference (RD) = 1.73, 95% CI 2-sided [-10.18 to 13.65], Standard Error of Mean 6.08
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.021, Normal approximation for two proportions; Risk Difference (RD) = 17.12, 95% CI 2-sided [2.56 to 31.68], Standard Error of Mean 7.43
Statistical Analysis 9: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.064, Normal approximation for two proportions; Risk Difference (RD) = 13.27, 95% CI 2-sided [-0.79 to 27.34], Standard Error of Mean 7.17
Statistical Analysis 10: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.292, Normal approximation for two proportions; Risk Difference (RD) = 7.47, 95% CI 2-sided [-6.42 to 21.36], Standard Error of Mean 7.09
Statistical Analysis 11: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.125, Normal approximation for two proportions; Risk Difference (RD) = 11.31, 95% CI 2-sided [-3.16 to 25.78], Standard Error of Mean 7.38
Statistical Analysis 12: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.078, Normal approximation for two proportions; Risk Difference (RD) = 13.24, 95% CI 2-sided [-1.49 to 27.96], Standard Error of Mean 7.51

12. Secondary Outcome: Percentage of Participants Achieving ASDAS Inactive Disease at Weeks 2, 4, 8 and 12
Description: The ASDAS inactive disease was calculated from the ASDAS data. The ASDAS inactive disease was defined as ASDAS <1.3 units. Missing data were handled by NRI/LOCF.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: FAS - n=number of responders at each visit
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 52 | 52 | 52 | 51
Percentage of participants
  Week 2 (n=1, 1, 1, 0) | 1.92 | 1.92 | 1.92 | 0.00
  Week 4 (n=1, 3, 4, 1) | 1.92 | 5.77 | 7.69 | 1.96
  Week 8 (n=3, 1, 5, 1) | 5.77 | 1.92 | 9.62 | 1.96
  Week 12 (n=7, 7, 8, 4) | 13.46 | 13.46 | 15.38 | 7.84
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.313, Normal approximation for two proportions; Risk Difference (RD) = 1.92, 95% CI 2-sided [-1.81 to 5.66], Standard Error of Mean 1.90
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.313, Normal approximation for two proportions; Risk Difference (RD) = 1.92, 95% CI 2-sided [-1.81 to 5.66], Standard Error of Mean 1.90
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.313, Normal approximation for two proportions; Risk Difference (RD) = 1.92, 95% CI 2-sided [-1.81 to 5.66], Standard Error of Mean 1.90
Statistical Analysis 4: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.989, Normal approximation for two proportions; Risk Difference (RD) = -0.04, 95% CI 2-sided [-5.37 to 5.29], Standard Error of Mean 2.72
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.313, Normal approximation for two proportions; Risk Difference (RD) = 3.81, 95% CI 2-sided [-3.58 to 11.20], Standard Error of Mean 3.77
Statistical Analysis 6: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.170, Normal approximation for two proportions; Risk Difference (RD) = 5.73, 95% CI 2-sided [-2.45 to 13.91], Standard Error of Mean 4.17
Statistical Analysis 7: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.313, Normal approximation for two proportions; Risk Difference (RD) = 3.81, 95% CI 2-sided [-3.58 to 11.20], Standard Error of Mean 3.77
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.989, Normal approximation for two proportions; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-5.37 to 5.29], Standard Error of Mean 2.72
Statistical Analysis 9: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.091, Normal approximation for two proportions; Risk Difference (RD) = 7.65, 95% CI 2-sided [-1.22 to 16.52], Standard Error of Mean 4.53
Statistical Analysis 10: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.353, Normal approximation for two proportions; Risk Difference (RD) = 5.62, 95% CI 2-sided [-6.23 to 17.47], Standard Error of Mean 6.05
Statistical Analysis 11: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.353, Normal approximation for two proportions; Risk Difference (RD) = 5.62, 95% CI 2-sided [-6.23 to 17.47], Standard Error of Mean 6.05
Statistical Analysis 12: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.228, Normal approximation for two proportions; Risk Difference (RD) = 7.54, 95% CI 2-sided [-4.73 to 19.81], Standard Error of Mean 6.26

13. Secondary Outcome: Change From Baseline in BASDAI Total Score at Week 2, 4, 8 and 12
Description: BASDAI is a validated self-assessment tool used to determine disease activity in participant with Ankylosing Spondylitis. Utilizing a Numerical Rating Scale (NRS) of 0-10 (0 = none and 10 = very severe) participant's answered 6 questions measuring discomfort, pain and fatigue. The BASDAI score is calculated by computing the mean of questions 5 and 6 and adding it to the sum of questions (Q)1-4. This score is then divided by 5. BASDAI=Q1+Q2+Q3+Q4+[Q5+Q6/2]/5. The final BASDAI score averages the individual assessments for a final score range of 0-10. Negative values indicate improvement.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 51 | 52 | 51 | 51
Units on a scale
  Week 2 | -1.45 (0.219) | -1.53 (0.217) | -1.24 (0.219) | -1.42 (0.219)
  Week 4 | -1.90 (0.242) | -1.93 (0.240) | -1.84 (0.242) | -1.60 (0.243)
  Week 8 | -2.16 (0.268) | -2.39 (0.267) | -2.35 (0.271) | -1.87 (0.271)
  Week 12 | -2.75 (0.277) | -2.88 (0.276) | -2.68 (0.281) | -1.85 (0.283)
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.926, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.64 to 0.58], Standard Error of Mean 0.310
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.718, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.72 to 0.50], Standard Error of Mean 0.308
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.570, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.43 to 0.79], Standard Error of Mean 0.310
Statistical Analysis 4: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.384, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.97 to 0.38], Standard Error of Mean 0.343
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.334, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-1.00 to 0.34], Standard Error of Mean 0.341
Statistical Analysis 6: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.474, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.92 to 0.43], Standard Error of Mean 0.343
Statistical Analysis 7: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.445, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-1.04 to 0.46], Standard Error of Mean 0.381
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.174, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-1.27 to 0.23], Standard Error of Mean 0.380
Statistical Analysis 9: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.217, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-1.23 to 0.28], Standard Error of Mean 0.383
Statistical Analysis 10: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.024, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.90, 95% CI 2-sided [-1.69 to -0.12], Standard Error of Mean 0.396
Statistical Analysis 11: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -1.03, 95% CI 2-sided [-1.81 to -0.24], Standard Error of Mean 0.396
Statistical Analysis 12: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.038, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.62 to -0.04], Standard Error of Mean 0.399

14. Secondary Outcome: Percentage of Participants Achieving a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)50 Response at Weeks 2, 4, 8 and 12
Description: BASDAI is a validated self-assessment tool used to determine disease activity in participant with Ankylosing Spondylitis. Utilizing a Numerical Rating Scale (NRS) of 0-10 (0 = none and 10 = very severe) participant's answered 6 questions measuring discomfort, pain and fatigue. The BASDAI score is calculated by computing the mean of questions 5 and 6 and adding it to the sum of questions (Q)1-4. This score is then divided by 5. The final BASDAI score range from 0-10. A positive response was defined as a 50% improvement in the BASDAI from baseline.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: FAS - n=number of responders at each visit
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 52 | 52 | 52 | 51
Percentage of participants
  Week 2 (n=6, 11, 7, 8) | 11.54 [2.92 to 20.61] | 21.15 | 13.46 | 15.69
  Week 4 (n=15, 12, 15, 11) | 28.85 | 23.08 | 28.85 | 21.57
  Week 8 (n=18, 17, 21, 14) | 34.62 | 32.69 | 40.38 | 27.45
  Week 12 (n=24, 22, 22, 12) | 46.15 | 42.31 | 42.31 | 23.53
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.539, Normal approximation for two proportions; Risk Difference (RD) = -4.15, 95% CI 2-sided [-17.38 to 9.08], Standard Error of Mean 6.75
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.473, Normal approximation for two proportions; Risk Difference (RD) = 5.47, 95% CI 2-sided [-9.46 to 20.40], Standard Error of Mean 7.62
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.749, Normal approximation for two proportions; Risk Difference (RD) = -2.22, 95% CI 2-sided [-15.85 to 11.40], Standard Error of Mean 6.95
Statistical Analysis 4: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.393, Normal approximation for two proportions; Risk Difference (RD) = 7.28, 95% CI 2-sided [-9.43 to 23.98], Standard Error of Mean 8.52
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.854, Normal approximation for two proportions; Risk Difference (RD) = 1.51, 95% CI 2-sided [-14.57 to 17.59], Standard Error of Mean 8.20
Statistical Analysis 6: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.393, Normal approximation for two proportions; Risk Difference (RD) = 7.28, 95% CI 2-sided [-9.43 to 23.98], Standard Error of Mean 8.52
Statistical Analysis 7: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.430, Normal approximation for two proportions; Risk Difference (RD) = 7.16, 95% CI 2-sided [-10.65 to 24.97], Standard Error of Mean 9.09
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.561, Normal approximation for two proportions; Risk Difference (RD) = 5.24, 95% CI 2-sided [-12.44 to 22.92], Standard Error of Mean 9.02
Statistical Analysis 9: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.162, Normal approximation for two proportions; Risk Difference (RD) = 12.93, 95% CI 2-sided [-5.17 to 31.04], Standard Error of Mean 9.24
Statistical Analysis 10: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.013, Normal approximation for two proportions; Risk Difference (RD) = 22.62, 95% CI 2-sided [4.76 to 40.49], Standard Error of Mean 9.11
Statistical Analysis 11: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.038, Normal approximation for two proportions; Risk Difference (RD) = 18.78, 95% CI 2-sided [1.01 to 36.55], Standard Error of Mean 9.07
Statistical Analysis 12: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.038, Normal approximation for two proportions; Risk Difference (RD) = 18.78, 95% CI 2-sided [1.01 to 36.55], Standard Error of Mean 9.07

15. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Weeks 2, 4, 8 and 12
Description: BASFI is a validated self-assessment tool that determines the degree of physical functional limitation in Ankylosing Spondylitis. Utilizing a Numerical Rating Scale (NRS) of 0-10 (0=easy, 10=impossible), participants answered 10 questions assessing their ability in completing normal daily activities or physically demanding activities. The BASFI score is a mean score of the 10 questions with lower scores indicating better physical function. The higher the negative value the better the improvement.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 51 | 52 | 51 | 51
Units on a scale
  Week 2 | -1.12 (0.192) | -1.16 (0.191) | -0.86 (0.192) | -0.74 (0.192)
  Week 4 | -1.36 (0.210) | -1.61 (0.208) | -1.32 (0.210) | -1.02 (0.210)
  Week 8 | -1.61 (0.247) | -2.07 (0.246) | -1.72 (0.249) | -1.38 (0.249)
  Week 12 | -1.90 (0.261) | -2.39 (0.260) | -2.24 (0.264) | -1.43 (0.266)
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.164, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.92 to 0.16], Standard Error of Mean 0.272
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.129, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.95 to 0.12], Standard Error of Mean 0.271
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.660, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.66 to 0.42], Standard Error of Mean 0.272
Statistical Analysis 4: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.256, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.92 to 0.25], Standard Error of Mean 0.297
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.048, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-1.17 to -0.00], Standard Error of Mean 0.296
Statistical Analysis 6: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.318, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.88 to 0.29], Standard Error of Mean 0.297
Statistical Analysis 7: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.522, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.92 to 0.47], Standard Error of Mean 0.350
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.050, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-1.38 to 0.00], Standard Error of Mean 0.350
Statistical Analysis 9: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.337, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-1.03 to 0.36], Standard Error of Mean 0.352
Statistical Analysis 10: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.214, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-1.20 to 0.27], Standard Error of Mean 0.373
Statistical Analysis 11: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-1.69 to -0.22], Standard Error of Mean 0.372
Statistical Analysis 12: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.031, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-1.55 to -0.08], Standard Error of Mean 0.375

16. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) at Weeks 2, 4, 8 and 12
Description: BASMI is an objective measure of spinal mobility and was completed by a blinded assessor. The BASMI score is composed of 5 clinical measures: cervical rotation, intermalleolar distance, modified Schober's test, lateral flexion and tragus to wall distance. The derived score used the average of the 5 assessments on a scale of 0-10 scale with higher scores indicating more impairment of spinal mobility. BASMI was analyzed using the linear function method. The higher the negative value the better the improvement.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 51 | 51 | 51 | 51
Units on a scale
  Week 2 | -0.09 (0.075) | -0.24 (0.075) | -0.22 (0.075) | -0.09 (0.075)
  Week 4 | -0.15 (0.083) | -0.24 (0.083) | -0.26 (0.084) | -0.14 (0.084)
  Week 8 | -0.34 (0.095) | -0.40 (0.095) | -0.48 (0.096) | -0.19 (0.096)
  Week 12 | -0.33 (0.109) | -0.42 (0.109) | -0.55 (0.111) | -0.16 (0.112)
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.982, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.21 to 0.21], Standard Error of Mean 0.106
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.151, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.36 to 0.06], Standard Error of Mean 0.106
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.205, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.34 to 0.07], Standard Error of Mean 0.106
Statistical Analysis 4: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.898, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.25 to 0.22], Standard Error of Mean 0.118
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.370, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.34 to 0.13], Standard Error of Mean 0.118
Statistical Analysis 6: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.288, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.36 to 0.11], Standard Error of Mean 0.119
Statistical Analysis 7: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.242, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.42 to 0.11], Standard Error of Mean 0.135
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.120, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.48 to 0.06], Standard Error of Mean 0.135
Statistical Analysis 9: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.031, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.56 to -0.03], Standard Error of Mean 0.136
Statistical Analysis 10: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.280, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.48 to 0.14], Standard Error of Mean 0.157
Statistical Analysis 11: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.099, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.57 to 0.05], Standard Error of Mean 0.157
Statistical Analysis 12: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.014, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.70 to -0.08], Standard Error of Mean 0.158

17. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) at Weeks 4, 8 and 12
Description: Assessment of enthesitis of 13 sites was performed in the following, 1st costochondral joint left and right, 7th costochondral joint left and right, posterior superior iliac spine left and right, anterior superior iliac spine left and right, iliac crest left and right, 5th lumbar spinous process and proximal insertion of Achilles tendon left and right. Each site was graded for the presence (1) and absence (0) of tenderness yielding total MASES ranging from 0 (no tenderness) to 13 (worst possible score; severe tenderness).
Time Frame: Baseline, Week 4, Week 8, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 51 | 51 | 50 | 50
Units on a scale
  Week 4 | -0.16 (0.272) | -0.93 (0.271) | -0.89 (0.274) | -0.11 (0.275)
  Week 8 | -0.79 (0.289) | -1.19 (0.289) | -0.97 (0.295) | -0.54 (0.292)
  Week 12 | -0.66 (0.259) | -1.37 (0.259) | -1.24 (0.263) | -0.34 (0.265)
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.895, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.81 to 0.71], Standard Error of Mean 0.387
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.033, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.59 to -0.07], Standard Error of Mean 0.386
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.044, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-1.55 to -0.02], Standard Error of Mean 0.388
Statistical Analysis 4: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.530, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-1.07 to 0.55], Standard Error of Mean 0.411
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.114, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-1.46 to 0.16], Standard Error of Mean 0.411
Statistical Analysis 6: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.297, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-1.25 to 0.38], Standard Error of Mean 0.415
Statistical Analysis 7: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.377, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-1.06 to 0.40], Standard Error of Mean 0.370
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -1.04, 95% CI 2-sided [-1.77 to -0.31], Standard Error of Mean 0.370
Statistical Analysis 9: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.017, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.90, 95% CI 2-sided [-1.64 to -0.17], Standard Error of Mean 0.373

18. Secondary Outcome: Extra-Articular Involvement From Specific Ankylosing Spondylitis Medical History
Description: Participants were assessed at Baseline, Week 12 and Week 16 (Follow-up) to determine if they had specific Ankylosing Spondylitis medical history or changes in specific Ankylosing Spondylitis medical history which included: Inflammatory Bowel Disease (IBD), Peripheral Articular Involvement (PAI; as assessed by swollen joint count), psoriasis (PSO) and uveitis (UVE).
Time Frame: Baseline, Week 12 and Follow-up
Population: FAS - n=number of participants completing the Specific Medical History Assessment at each visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 6 | 9 | 6 | 4
Percentage of Participants
  IBD: Never: Baseline (n=6, 9, 6, 4) | 100 | 88.9 | 100 | 100
  IBD: Past But Not Active: Baseline (n=6, 9, 6, 4) | 0 | 0 | 0 | 0
  IBD: Currently Active: Baseline (n=6, 9, 6, 4) | 0 | 11.1 | 0 | 0
  IBD: New Condition: Baseline (n=6, 9, 6, 4) | 0 | 0 | 0 | 0
  IBD: Never: Week 4 (n=4, 7, 3, 2) | 100 | 100 | 100 | 100
  IBD: Past But Not Active: Week 4 (n=4, 7, 3, 2) | 0 | 0 | 0 | 0
  IBD: Currently Active: Week 4 (n=4, 7, 3, 2) | 0 | 0 | 0 | 0
  IBD: New Condition: Week 4 (n=4, 7, 3, 2) | 0 | 0 | 0 | 0
  IBD: Never: Week 8 (n=2, 6, 2, 4) | 100 | 100 | 100 | 100
  IBD: Past But Not Active: Week 8 (n=2, 6, 2, 4) | 0 | 0 | 0 | 0
  IBD: Currently Active: Week 8 (n=2, 6, 2, 4) | 0 | 0 | 0 | 0
  IBD: New Condition: Week 8 (n=2, 6, 2, 4) | 0 | 0 | 0 | 0
  IBD: Never: Week 12 (n=5, 6, 2, 3) | 100 | 100 | 100 | 100
  IBD: Past But Not Active: Week 12 (n=5, 6, 2, 3) | 0 | 0 | 0 | 0
  IBD: Currently Active: Week 12 (n=5, 6, 2, 3) | 0 | 0 | 0 | 0
  IBD: New Condition: Week 12 (n=5, 6, 2, 3) | 0 | 0 | 0 | 0
  IBD: Never: Follow-up (n=3, 6, 4, 2) | 100 | 100 | 100 | 100
  IBD: Past But Not Active: Follow-up (n=3, 6, 4, 2) | 0 | 0 | 0 | 0
  IBD: Currently Active: Follow-up (n=3, 6, 4, 2) | 0 | 0 | 0 | 0
  IBD: New Condition: Follow-up (n=3, 6, 4, 2) | 0 | 0 | 0 | 0
  PAI: Never: Baseline (n=6, 9, 6, 4) | 33.3 | 44.4 | 0 | 25.0
  PAI: Past But Not Active: Baseline (n=6, 9, 6, 4) | 0 | 0 | 16.7 | 0
  PAI: Currently Active: Baseline (n=6, 9, 6, 4) | 66.7 | 44.4 | 66.7 | 75.0
  PAI: New condition: Baseline (n=6, 9, 6, 4) | 0 | 11.1 | 16.7 | 0
  PAI: Never: Week 4 (n=4, 7, 3, 2) | 0 | 28.6 | 0 | 0
  PAI: Past But Not Active: Week 4 (n=4, 7, 3, 2) | 0 | 14.3 | 33.3 | 0
  PAI: Currently Active: Week 4 (n=4, 7, 3, 2) | 100 | 57.1 | 66.7 | 100
  PAI: New condition: Week 4 (n=4, 7, 3, 2) | 0 | 0 | 0 | 0
  PAI: Never: Week 8 (n=2, 6, 2, 4) | 0 | 50.0 | 0 | 0
  PAI: Past But Not Active: Week 8 (n=2, 6, 2, 4) | 0 | 0 | 50.0 | 0
  PAI: Currently Active: Week 8 (n=2, 6, 2, 4) | 100 | 50.0 | 50.0 | 100
  PAI: New Condition: Week 8 (n=2, 6, 2, 4) | 0 | 0 | 0 | 0
  PAI: Never: Week 12 (n=5, 5, 2, 3) | 20.0 | 40.0 | 0 | 0
  PAI: Past But Not Active: Week 12 (n=5, 5, 2, 3) | 0 | 0 | 0 | 0
  PAI: Currently Active: Week 12 (n=5, 5, 2, 3) | 40.0 | 60.0 | 100 | 100
  PAI: New Condition: Week 12 (n=5, 5, 2, 3) | 40.0 | 0 | 0 | 0
  PAI: Never: Follow-up (n=3, 6, 4, 2) | 0 | 50.0 | 25.0 | 0
  PAI: Past But Not Active: Follow-up (n=3, 6, 4, 2) | 0 | 0 | 25.0 | 0
  PAI: Currently Active: Follow-up (n=3, 6, 4, 2) | 66.7 | 50.0 | 50.0 | 100
  PAI: New Condition: Follow-up (n=3, 6, 4, 2) | 33.3 | 0 | 0 | 0
  PSO: Never: Baseline (n=6, 9, 6, 4) | 100 | 88.9 | 83.3 | 75.0
  PSO: Past But Not Active: Baseline (n=6, 9, 6, 4) | 0 | 0 | 0 | 0
  PSO: Currently Active: Baseline (n=6, 9, 6, 4) | 0 | 11.1 | 16.7 | 25.0
  PSO: New Condition: Baseline (n=6, 9, 6, 4) | 0 | 0 | 0 | 0
  PSO: Never: Week 4 (n=4, 7, 3, 2) | 100 | 85.7 | 66.7 | 100
  PSO: Past But Not Active: Week 4 (n=4, 7, 3, 2) | 0 | 0 | 0 | 0
  PSO: Currently Active: Week 4 (n=4, 7, 3, 2) | 0 | 14.3 | 33.3 | 0
  PSO: New Condition: Week 4 (n=4, 7, 3, 2) | 0 | 0 | 0 | 0
  PSO: Never: Week 8 (n=2, 6, 2, 4) | 100 | 83.3 | 50.0 | 100
  PSO: Past But Not Active: Week 8 (n=2, 6, 2, 4) | 0 | 0 | 0 | 0
  PSO: Currently Active: Week 8 (n=2, 6, 2, 4) | 0 | 16.7 | 50.0 | 0
  PSO: New Condition: Week 8 (n=2, 6, 2, 4) | 0 | 0 | 0 | 0
  PSO: Never: Week 12 (n=5, 6, 2, 3) | 80.0 | 83.3 | 100 | 100
  PSO: Past But Not Active: Week 12 (n=5, 6, 2, 3) | 20.0 | 0 | 0 | 0
  PSO: Currently Active: Week 12 (n=5, 6, 2, 3) | 0 | 16.7 | 0 | 0
  PSO: New Condition: Week 12 (n=5, 6, 2, 3) | 0 | 0 | 0 | 0
  PSO: Never: Follow-up (n=3, 6, 4, 2) | 100 | 83.3 | 100 | 100
  PSO: Past But Not Active: Follow-up (n=3, 6, 4, 2) | 0 | 0 | 0 | 0
  PSO: Currently Active: Follow-up (n=3, 6, 4, 2) | 0 | 16.7 | 0 | 0
  PSO: New Condition: Follow-up (n=3, 6, 4, 2) | 0 | 0 | 0 | 0
  UVE: Never: Baseline (n=6, 9, 6, 4) | 50.0 | 55.6 | 83.3 | 100
  UVE: Past But Not Active: Baseline (n=6, 9, 6, 4) | 16.7 | 33.3 | 0 | 0
  UVE: Currently Active: Baseline (n=6, 9, 6, 4) | 33.3 | 11.1 | 16.7 | 0
  UVE: New Condition: Baseline (n=6, 9, 6, 4) | 0 | 0 | 0 | 0
  UVE: Never: Week 4 (n=4, 7, 3, 2) | 75.0 | 71.4 | 66.7 | 100
  UVE: Past But Not Active: Week 4 (n=4, 7, 3, 2) | 25.0 | 28.6 | 33.3 | 0
  UVE: Currently Active: Week 4 (n=4, 7, 3, 2) | 0 | 0 | 0 | 0
  UVE: New Condition: Week 4 (n=4, 7, 3, 2) | 0 | 0 | 0 | 0
  UVE: Never: Week 8 (n=2, 6, 2, 4) | 100 | 50.0 | 50.0 | 100
  UVE: Past But Not Active: Week 8 (n=2, 6, 2, 4) | 0 | 50.0 | 50.0 | 0
  UVE: Currenly Active: Week 8 (n=2, 6, 2, 4) | 0 | 0 | 0 | 0
  UVE: New Condition: Week 8 (n=2, 6, 2, 4) | 0 | 0 | 0 | 0
  UVE: Never: Week 12 (n=5, 6, 2, 3) | 40.0 | 66.7 | 50.0 | 100
  UVE: Past But Not Active: Week 12 (n=5, 6, 2, 3) | 60.0 | 33.3 | 50.0 | 0
  UVE: Currently Active: Week 12 (n=5, 6, 2, 3) | 0 | 0 | 0 | 0
  UVE: New Condition: Week 12 (n=5, 6, 2, 3) | 0 | 0 | 0 | 0
  UVE: Never: Follow-up (n=3, 6, 4, 2) | 100 | 50.0 | 50.0 | 100
  UVE: Past But Not Active: Follow-up (n=3, 6, 4, 2) | 0 | 33.3 | 25.0 | 0
  UVE: Currently Active: Follow-up (n=3, 6, 4, 2) | 0 | 16.7 | 0 | 0
  UVE: New Condition: Follow-up (n=3, 6, 4, 2) | 0 | 0 | 25.0 | 0

19. Secondary Outcome: Change From Baseline of Total Swollen Joint Count at Weeks 2, 4 8 and 12
Description: This assessment was performed by the blinded assessor using the following scale: Present/Absent/Not Done/Not Applicable (to be used for artificial or missing joints) for determination of the total number of swollen joints. Forty-four joints were assessed for swelling on left and right side and included the following: sternoclaviculars, acromioclaviculars, shoulders, elbows, wrists, metacarpophalangeals (I, II, III, IV, V), thumb interphalangeal, proximal interphalangeals (II, III, IV, V), knees, ankles, and metatarsophalangeals (I, II, III, IV, V). Artificial joints were not assessed. A negative change means improvement.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Swollen Joints
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 51 | 52 | 51 | 51
Swollen Joints
  Week 2 | -0.53 (0.293) | 0.23 (0.291) | -1.20 (0.292) | -0.43 (0.293)
  Week 4 | -0.87 (0.260) | -0.57 (0.259) | -1.23 (0.260) | -0.86 (0.261)
  Week 8 | -1.02 (0.442) | -0.98 (0.442) | -1.28 (0.451) | -0.60 (0.448)
  Week 12 | -0.87 (0.362) | -0.79 (0.362) | -1.40 (0.368) | -0.99 (0.373)
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.800, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.92 to 0.71], Standard Error of Mean 0.414
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.113, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [-0.16 to 1.47], Standard Error of Mean 0.413
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.064, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-1.59 to 0.05], Standard Error of Mean 0.414
Statistical Analysis 4: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.972, Mixed Models Analysis; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.74 to 0.71], Standard Error of Mean 0.368
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.440, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.44 to 1.01], Standard Error of Mean 0.368
Statistical Analysis 6: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.311, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-1.10 to 0.35], Standard Error of Mean 0.369
Statistical Analysis 7: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.501, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.66 to 0.82], Standard Error of Mean 0.629
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.543, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-1.63 to 0.86], Standard Error of Mean 0.629
Statistical Analysis 9: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.287, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-1.93 to 0.57], Standard Error of Mean 0.636
Statistical Analysis 10: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.820, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.91 to 1.14], Standard Error of Mean 0.519
Statistical Analysis 11: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.711, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.83 to 1.22], Standard Error of Mean 0.520
Statistical Analysis 12: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.424, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.45 to 0.61], Standard Error of Mean 0.524

20. Secondary Outcome: Change From Baseline of Mean Spinal Mobility (Chest Expansion) at Week 2, 4, 8 and 12
Description: Chest expansion, measured in centimeters (cm), is defined as the difference in the thoracic circumference during full expiration versus full inspiration. This was measured at the 4th intercostal space. The difference between maximal inspiration and expiration of the two attempts was recorded. The better of the two attempts was used to calculate chest expansion. Missing data at Week 12 were imputed by LOCF if data at an early visit (discontinuation visit) were available.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 51 | 51 | 51 | 51
cm
  Week 2 | 0.30 (0.144) | 0.35 (0.143) | -0.03 (0.144) | 0.24 (0.144)
  Week 4 | 0.54 (0.164) | 0.13 (0.162) | 0.13 (0.164) | 0.38 (0.165)
  Week 8 | 0.52 (0.178) | 0.35 (0.178) | 0.15 (0.182) | 0.13 (0.181)
  Week 12 | 0.69 (0.187) | 0.49 (0.187) | 0.13 (0.190) | 0.31 (0.193)
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.785, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.34 to 0.46], Standard Error of Mean 0.203
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.605, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.30 to 0.51], Standard Error of Mean 0.203
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.175, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.68 to 0.12], Standard Error of Mean 0.204
Statistical Analysis 4: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.482, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.29 to 0.62], Standard Error of Mean 0.232
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.288, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.70 to 0.21], Standard Error of Mean 0.231
Statistical Analysis 6: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.278, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.71 to 0.21], Standard Error of Mean 0.233
Statistical Analysis 7: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.134, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-0.12 to 0.88], Standard Error of Mean 0.254
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.397, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.29 to 0.72], Standard Error of Mean 0.254
Statistical Analysis 9: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.964, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.50 to 0.52], Standard Error of Mean 0.257
Statistical Analysis 10: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.155, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-0.15 to 0.91], Standard Error of Mean 0.269
Statistical Analysis 11: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.491, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.34 to 0.72], Standard Error of Mean 0.269
Statistical Analysis 12: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.515, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.71 to 0.36], Standard Error of Mean 0.271

21. Secondary Outcome: Change From Baseline to Week 12 in Short-Form-36 Health Survey (SF-36) Physical and Mental Health Scores at Week 12
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and wellbeing: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (0=no functioning, 100=highest level of functioning). Missing data at Week 12 were imputed by LOCF if data at an early visit (discontinuation visit) were available.
Time Frame: Baseline, Week 12
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 52 | 52 | 52 | 51
Units on a scale
  Week 12 Physical Health Score | 6.34 (0.923) | 6.49 (0.914) | 7.05 (0.943) | 2.69 (0.932)
  Week 12 Mental Health Score | 2.08 (1.306) | 4.15 (1.294) | 3.71 (1.336) | 2.41 (1.318)
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Physical Health Score; Test type: Superiority or Other; p = 0.006, ANCOVA; ANCOVA model includes fixed effects for treatment group and baseline value as a covariate; Mean Difference (Final Values) = 3.65, 95% CI 2-sided [1.06 to 6.24], Standard Error of Mean 1.312
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Physical Health Score; Test type: Superiority or Other; p = 0.004, ANCOVA; ANCOVA model includes fixed effects for treatment group and baseline value as a covariate; Mean Difference (Final Values) = 3.80, 95% CI 2-sided [1.23 to 6.37], Standard Error of Mean 1.305
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Physical Health Score; Test type: Superiority or Other; p = 0.001, ANCOVA; ANCOVA model includes fixed effects for treatment group and baseline value as a covariate; Mean Difference (Final Values) = 4.36, 95% CI 2-sided [1.74 to 6.98], Standard Error of Mean 1.328
Statistical Analysis 4: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Mental Health Score; Test type: Superiority or Other; p = 0.857, ANCOVA; ANCOVA model includes fixed effects for treatment group and baseline value as a covariate; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-4.00 to 3.33], Standard Error of Mean 1.857
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Mental Health Score; Test type: Superiority or Other; p = 0.350, ANCOVA; ANCOVA model includes fixed effects for treatment group and baseline value as a covariate; Mean Difference (Final Values) = 1.73, 95% CI 2-sided [-1.91 to 5.37], Standard Error of Mean 1.848
Statistical Analysis 6: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Mental Health Score; Test type: Superiority or Other; p = 0.490, ANCOVA; ANCOVA model includes fixed effects for treatment group and baseline value as a covariate; Mean Difference (Final Values) = 1.30, 95% CI 2-sided [-2.40 to 5.00], Standard Error of Mean 1.876

22. Secondary Outcome: Change From Baseline in EuroQol EQ-5D Health State Profile (EQ-5D) Utility Score at Week 12
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of single utility score. Health state profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression; Scale range 1 to 3 (1=better health state [no problems], 3=worst health state [confined to bed]).
Time Frame: Baseline, Week 12
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 52 | 52 | 52 | 51
Units on a scale | 0.17 (0.034) | 0.16 (0.034) | 0.22 (0.035) | 0.10 (0.034)
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.125, ANCOVA; ANCOVA model includes fixed effects for treatment group and baseline value as a covariate; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.02 to 0.17], Standard Error of Mean 0.048
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.207, ANCOVA; ANCOVA model includes fixed effects for treatment group and baseline value as a covariate; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.03 to 0.16], Standard Error of Mean 0.048
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.013, ANCOVA; ANCOVA model includes fixed effects for treatment group and baseline value as a covariate; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [0.03 to 0.22], Standard Error of Mean 0.049

23. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score at Weeks 2, 4, 8 and 12
Description: FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (not at all) to 4 (very much). Larger the participant's response to the questions (with the exception of 2 negatively stated), greater was the participant's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score).
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 51 | 51 | 51 | 51
Units on a scale
  Week 2 | 3.62 (0.871) | 1.97 (0.871) | 2.17 (0.875) | 1.90 (0.872)
  Week 4 | 4.25 (0.931) | 3.67 (0.927) | 2.80 (0.937) | 2.71 (0.938)
  Week 8 | 4.54 (1.039) | 4.81 (1.039) | 4.19 (1.061) | 2.85 (1.053)
  Week 12 | 4.74 (1.145) | 7.03 (1.145) | 7.58 (1.166) | 3.08 (1.178)
Statistical Analysis 1: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.163, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.72, 95% CI 2-sided [-0.71 to 4.15], Standard Error of Mean 1.232
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.955, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-2.36 to 2.50], Standard Error of Mean 1.232
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 2; Test type: Superiority or Other; p = 0.826, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-2.17 to 2.71], Standard Error of Mean 1.237
Statistical Analysis 4: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.246, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.54, 95% CI 2-sided [-1.07 to 4.14], Standard Error of Mean 1.322
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.467, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.96, 95% CI 2-sided [-1.64 to 3.56], Standard Error of Mean 1.318
Statistical Analysis 6: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 4; Test type: Superiority or Other; p = 0.948, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-2.53 to 2.70], Standard Error of Mean 1.328
Statistical Analysis 7: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.255, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.69, 95% CI 2-sided [-1.23 to 4.61], Standard Error of Mean 1.479
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.187, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.96, 95% CI 2-sided [-0.96 to 4.87], Standard Error of Mean 1.479
Statistical Analysis 9: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 8; Test type: Superiority or Other; p = 0.373, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.34, 95% CI 2-sided [-1.62 to 4.29], Standard Error of Mean 1.497
Statistical Analysis 10: Comparison: Tofacitinib 2 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.313, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.66, 95% CI 2-sided [-1.58 to 4.90], Standard Error of Mean 1.643
Statistical Analysis 11: Comparison: Tofacitinib 5 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.017, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 3.95, 95% CI 2-sided [0.71 to 7.19], Standard Error of Mean 1.642
Statistical Analysis 12: Comparison: Tofacitinib 10 mg BID vs Placebo BID; Week 12; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 4.51, 95% CI 2-sided [1.23 to 7.78], Standard Error of Mean 1.660

ADVERSE EVENTS:
Time Frame: From informed consent through and including 28 calendar days after the last administration of the investigational product.
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Tofacitinib 2 mg BID | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo BID
Serious Adverse Events (participants affected / at risk) | 0/52 | 1/52 | 1/52 | 2/51
Other Adverse Events (participants affected / at risk) | 15/52 | 10/52 | 13/52 | 14/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Tofacitinib 2 mg BID (N=52) | Tofacitinib 5 mg BID (N=52) | Tofacitinib 10 mg BID (N=52) | Placebo BID (N=51)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Iridocyclitis (Eye disorders) | 0 | 1 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0/18 | 0/13 | 0/14 | 1/19
Uterine spasm (Reproductive system and breast disorders) | 0/18 | 0/13 | 0/14 | 1/19
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/18 | 0/13 | 0/14 | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Tofacitinib 2 mg BID (N=52) | Tofacitinib 5 mg BID (N=52) | Tofacitinib 10 mg BID (N=52) | Placebo BID (N=51)
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 4 | 4 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 3 | 1
Vaginitis bacterial (Infections and infestations) | 0/18 | 0/13 | 0/14 | 1/19
Vulvovaginal mycotic infection (Infections and infestations) | 1/18 | 0/13 | 0/14 | 0/19
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 2 | 2 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/18 | 0/13 | 0/14 | 1/19
Haematuria (Renal and urinary disorders) | 0 | 1 | 2 | 1
Balanoposthitis (Reproductive system and breast disorders) | 1/34 | 0/39 | 0/38 | 0/32
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less